CLINICAL TRIAL: NCT04933643
Title: Analysis of Influencing Factors of Gastric Preparation Quality for Magnetically Controlled Capsule Gastroscopy
Brief Title: Analysis of Influencing Factors of Gastric Preparation Quality for MCCG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Other Study IDs: 2020SDU-QILU-072
Record Dates: First submitted 2021-05-19; First posted 2021-06-22 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Capsule Endoscopy
Keywords: Magnetically Controlled Capsule Gastroscopy; Influencing Factors; Gastric Preparation Quality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- well prepared: GCS was the total scores of all six land-marks, ranging from 6 (completely unprepared) to 24 (perfect). We define that the stomach is well prepared when GCS ≥ 18
- inadequate prepared: GCS was the total scores of all six land-marks, ranging from 6 (completely unprepared) to 24 (perfect). We define that GCS < 18 is inadequate.

INTERVENTIONS:
Other:

SUMMARY:
The invention of magnetically controlled capsule gastroscopy makes the movement of capsule endoscope in the body controllable. Endoscopic doctors can adjust the angle of capsule observation to examine gastric mucosa according to the need of examination. However, The presence of food residue, air bubbles, mucus and bile in the gastric cavity will affect the observation of gastric mucosa by capsule endoscopy. it will reduce the completion rate of capsule endoscopy, and even lead to misdiagnosis and missed diagnosis. The purpose of this study is to explore the factors affecting the quality of gastroscopy gastric environmental preparation of magnetically capsule.

DETAILED DESCRIPTION:
Magnetically controlled capsule endoscopy is different from ordinary electronic gastroenteroscopy, it can not fill and clean the gastric cavity by water injection. The presence of food residue, air bubbles, mucus and bile in the gastric cavity will affect the observation of gastric mucosa by capsule endoscopy, reduce the completion rate of capsule endoscopy, and even lead to misdiagnosis and missed diagnosis, so the quality of MCCG gastric environmental preparation is an important factor limiting the accuracy of diagnosis of gastric lesions. We design the case report table by consulting the literature, and then collect patient information, and speculate the relevant influencing factors through the evaluation of the quality of gastric environmental preparation of the examination results. the ultimate goal is to reduce the missed diagnosis rate and misdiagnosis rate and the waste of clinical resources, to prepare the gastric environment more pertinently, and to provide certain guiding significance for the preparation of gastric environment in clinical magnetically controlled capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-75 years old who intend to undergo magnetron capsule gastroscopy, regardless of gender
* sign informed consent form

Exclusion Criteria:

* dysphagia, known or suspected gastrointestinal obstruction、stricture and fistula
* patients with severe somatic diseases unable to complete examination
* known active upper gastrointestinal bleeding
* previous history of upper digestive tract or abdominal surgery to change
* gastrointestinal anatomy
* patients with cardiac pacemakers or implanted with other electronic medical
* instruments and magnetic metal foreign bodies
* pregnant women
* claustrophobia or other mental disorders uncontrollable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged 18-75 years old who intend to undergo magnetron capsule gastroscopy, regardless of gender
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
GCS score was used to evaluate the quality of gastric preparation | 24 months
  GCS score was used to evaluate the quality of gastric preparation. GCS was defined as the sum of the scores of six major anatomical markers of the stomach (heart, fundus, body, horn, sinus, and pylorus).A 4-point grading system was used to define cleanliness as excellent (no mucus and foam attachment :4 points);Good (there is a small amount of mucus and foam, but it does not affect the test: score 3 points);Average (with a fair amount of mucus or foam).Failure to complete a completely reliable examination :2 points);Poor (large amount of mucus or foam residue :1 point).The GCS is the total score for all six landmarks, ranging from 6 (completely unprepared) to 24 (perfect).Gastric preparation was defined as sufficient when GCS≥18 and insufficient when GCS<18.
Questionnaire data were used to analyze the influencing factors | 24 months
  Before the examination, the subjects were required to fill in a questionnaire about the influencing factors of the quality of stomach preparation. According to GCS, the subjects were divided into fully prepared group and inadequately prepared group. Finally, statistical analysis was used to find the influencing factors that had statistical significance with the quality of stomach preparation according to the questionnaire content.

SECONDARY OUTCOMES:
The number of positive lesions | 24 months
  The positive lesions detected in this study refer to some focal lesions of the stomach, including polyps, ulcers, gastric varices, submucosal tumors and so on.The lesions were identified by physicians who had performed magnetic capsule gastroscopy in more than 400 cases.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months
  The safety of MCCG includes the acceptability or adverse events of MCCG preparation and examination, which is defined as symptoms or signs such as drinking water, examination and swallowing capsules, such as monitoring abdominal distension, nausea or vomiting.we count the number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China